CLINICAL TRIAL: NCT00435773
Title: Single and Repeated Leech Therapy for the Treatment of Late Stage Knee Osteoarthritis. A Randomized, Placebo Controlled Comparative Trial
Brief Title: Leeches for the Treatment of Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: University Hospital, Aachen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EK 102/03
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Last update posted 2007-04-09 (Estimated); Status verified 2007-04

CONDITIONS: Osteoarthritis; Arthralgia
Keywords: Osteoarthritis; Leeching; Randomized Controlled Trial; Arthralgia
MeSH Terms: conditions — Osteoarthritis; Arthralgia | interventions — Leeching

INTERVENTIONS:
Procedure: Single Leeching
Procedure: Repeated Leeching after 4 weeks
Procedure: Placebo Leeching

SUMMARY:
Previous studies have not addressed the question, whether or not a repeated leeching can supply symptomatic relief of osteoarthritic pain for extended periods of time. We present a randomized study to the effectiveness of single and repeated leech therapy in cases with advanced osteoarthritis of the knee using a large patient group compared to a control group, who were both blinded to the actual treatment modality.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of the knee
* Persistent osteoarthritic symptoms for at least 6 months
* Radiographic evidence of late stage osteoarthritis of the knee (stage III-IV)
* History of conservative management including pain medication and physical therapy

Exclusion Criteria:

* Anticoagulant treatment or history of hemophilia
* History or presence of rheumatic diseases leading to secondary osteoarthritis
* Presence of hematological, hepatic, renal or immunological disease
* Insulin-dependant diabetes mellitus
* Intraarticular injections or systemic application of corticosteroids during the 3 preceding months
* History of surgery of the affected knee during the last 3 months or joint replacement
* History of previous leech therapy
* Lack of informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118
Dates: Start 2004-02; Study Completion 2004-12

PRIMARY OUTCOMES:
KOOS Score overall (Clinical score)before intervention, after 1,4 and 6 weeks, 3 and 6 months
WOMAC Score overall (Clinical score)before intervention, after 1,4 and 6 weeks, 3 and 6 months
VAS (Visual analog scale, pain score)before intervention, after 1,4 and 6 weeks, 3 and 6 months

SECONDARY OUTCOMES:
KOOS subscores before intervention, after 1,4 and 6 weeks, 3 and 6 months
WOMAC subscores before intervention, after 1,4 and 6 weeks, 3 and 6 months
Requirement of pain medication before intervention, after 1,4 and 6 weeks, 3 and 6 months
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Andereya, MD, Study Chair — Department of Orthopaedic Surgery, University Hospital of the RWTH Aachen, Germany
Locations (1):
- Department of Orthopaedic Surgery, University Hospital of the RWTH Aachen, Germany, Aachen, Germany

REFERENCES:
- [Background] Hyson JM. Leech therapy: a history. J Hist Dent. 2005 Mar;53(1):25-7. PMID 15926663
- [Background] Whitaker IS, Izadi D, Oliver DW, Monteath G, Butler PE. Hirudo Medicinalis and the plastic surgeon. Br J Plast Surg. 2004 Jun;57(4):348-53. doi: 10.1016/j.bjps.2003.12.016. PMID 15145739
- [Background] Rao J, Whitaker IS. Use of Hirudo medicinalis by maxillofacial surgical units in the United Kingdom: current views and practice. Br J Oral Maxillofac Surg. 2003 Feb;41(1):54-5. doi: 10.1016/s0266-4356(02)00284-x. No abstract available. PMID 12576043
- [Background] Weinfeld AB, Yuksel E, Boutros S, Gura DH, Akyurek M, Friedman JD. Clinical and scientific considerations in leech therapy for the management of acute venous congestion: an updated review. Ann Plast Surg. 2000 Aug;45(2):207-12. doi: 10.1097/00000637-200045020-00021. PMID 10949353
- [Background] Dabb RW, Malone JM, Leverett LC. The use of medicinal leeches in the salvage of flaps with venous congestion. Ann Plast Surg. 1992 Sep;29(3):250-6. doi: 10.1097/00000637-199209000-00010. PMID 1524375
- [Background] Hayden RE, Phillips JG, McLear PW. Leeches. Objective monitoring of altered perfusion in congested flaps. Arch Otolaryngol Head Neck Surg. 1988 Dec;114(12):1395-9. doi: 10.1001/archotol.1988.01860240045021. PMID 3190866
- [Background] Hernandez-Diaz S, Varas-Lorenzo C, Garcia Rodriguez LA. Non-steroidal antiinflammatory drugs and the risk of acute myocardial infarction. Basic Clin Pharmacol Toxicol. 2006 Mar;98(3):266-74. doi: 10.1111/j.1742-7843.2006.pto_302.x. PMID 16611201
- [Background] Hernandez-Diaz S, Garcia-Rodriguez LA. Epidemiologic assessment of the safety of conventional nonsteroidal anti-inflammatory drugs. Am J Med. 2001 Feb 19;110 Suppl 3A:20S-7S. doi: 10.1016/s0002-9343(00)00682-3. PMID 11173046
- [Background] Pilcher H. Medicinal leeches: stuck on you. Nature. 2004 Nov 4;432(7013):10-1. doi: 10.1038/432010a. No abstract available. PMID 15525954
- [Background] Michalsen A, Moebus S, Spahn G, Esch T, Langhorst J, Dobos GJ. Leech therapy for symptomatic treatment of knee osteoarthritis: results and implications of a pilot study. Altern Ther Health Med. 2002 Sep-Oct;8(5):84-8. PMID 12233807
- [Background] Michalsen A, Klotz S, Ludtke R, Moebus S, Spahn G, Dobos GJ. Effectiveness of leech therapy in osteoarthritis of the knee: a randomized, controlled trial. Ann Intern Med. 2003 Nov 4;139(9):724-30. doi: 10.7326/0003-4819-139-9-200311040-00006. PMID 14597456
- [Background] Hochberg MC. Multidisciplinary integrative approach to treating knee pain in patients with osteoarthritis. Ann Intern Med. 2003 Nov 4;139(9):781-3. doi: 10.7326/0003-4819-139-9-200311040-00013. No abstract available. PMID 14597463
- [Background] Guyatt GH, Sackett DL, Cook DJ. Users' guides to the medical literature. II. How to use an article about therapy or prevention. A. Are the results of the study valid? Evidence-Based Medicine Working Group. JAMA. 1993 Dec 1;270(21):2598-601. doi: 10.1001/jama.270.21.2598. No abstract available. PMID 8230645
- [Background] Wolfe F, Lane NE. The longterm outcome of osteoarthritis: rates and predictors of joint space narrowing in symptomatic patients with knee osteoarthritis. J Rheumatol. 2002 Jan;29(1):139-46. PMID 11824950
- [Background] Hochberg MC, Altman RD, Brandt KD, Moskowitz RW. Design and conduct of clinical trials in osteoarthritis: preliminary recommendations from a task force of the Osteoarthritis Research Society. J Rheumatol. 1997 Apr;24(4):792-4. PMID 9101520
- [Background] Altman R, Brandt K, Hochberg M, Moskowitz R, Bellamy N, Bloch DA, Buckwalter J, Dougados M, Ehrlich G, Lequesne M, Lohmander S, Murphy WA Jr, Rosario-Jansen T, Schwartz B, Trippel S. Design and conduct of clinical trials in patients with osteoarthritis: recommendations from a task force of the Osteoarthritis Research Society. Results from a workshop. Osteoarthritis Cartilage. 1996 Dec;4(4):217-43. doi: 10.1016/s1063-4584(05)80101-3. No abstract available. PMID 11048620
- [Background] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Background] Roos EM, Klassbo M, Lohmander LS. WOMAC osteoarthritis index. Reliability, validity, and responsiveness in patients with arthroscopically assessed osteoarthritis. Western Ontario and MacMaster Universities. Scand J Rheumatol. 1999;28(4):210-5. doi: 10.1080/03009749950155562. PMID 10503556
- [Background] Whitaker IS, Rao J, Izadi D, Butler PE. Historical Article: Hirudo medicinalis: ancient origins of, and trends in the use of medicinal leeches throughout history. Br J Oral Maxillofac Surg. 2004 Apr;42(2):133-7. doi: 10.1016/S0266-4356(03)00242-0. PMID 15013545
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Lahav A, Burks RT, Greis PE, Chapman AW, Ford GM, Fink BP. Clinical outcomes following osteochondral autologous transplantation (OATS). J Knee Surg. 2006 Jul;19(3):169-73. doi: 10.1055/s-0030-1248101. PMID 16893154
- [Background] Englund M, Lohmander LS. Patellofemoral osteoarthritis coexistent with tibiofemoral osteoarthritis in a meniscectomy population. Ann Rheum Dis. 2005 Dec;64(12):1721-6. doi: 10.1136/ard.2005.035568. Epub 2005 Apr 20. PMID 15843446
- [Background] Kessler S, Lang S, Puhl W, Stove J. [The Knee Injury and Osteoarthritis Outcome Score--a multifunctional questionnaire to measure outcome in knee arthroplasty]. Z Orthop Ihre Grenzgeb. 2003 May-Jun;141(3):277-82. doi: 10.1055/s-2003-40083. German. PMID 12822074
- [Background] Markwardt F, Hauptmann J, Nowak G, Klessen C, Walsmann P. Pharmacological studies on the antithrombotic action of hirudin in experimental animals. Thromb Haemost. 1982 Jun 28;47(3):226-9. PMID 7112494
- [Background] Brown JE, Baugh RF, Hougie C. The inhibition of the intrinsic generation of activated factor X by heparin and hirudin. Thromb Res. 1980 Jan 1-15;17(1-2):267-72. doi: 10.1016/0049-3848(80)90314-x. No abstract available. PMID 7376133
- [Background] Dippenaar R, Smith J, Goussard P, Walters E. Meningococcal purpura fulminans treated with medicinal leeches. Pediatr Crit Care Med. 2006 Sep;7(5):476-8. doi: 10.1097/01.PCC.0000235422.23812.B4. PMID 16878049
- [Background] Ascenzi P, Amiconi G, Bode W, Bolognesi M, Coletta M, Menegatti E. Proteinase inhibitors from the European medicinal leech Hirudo medicinalis: structural, functional and biomedical aspects. Mol Aspects Med. 1995;16(3):215-313. doi: 10.1016/0098-2997(95)00002-x. No abstract available. PMID 8569452
- [Background] Rigbi M, Levy H, Eldor A, Iraqi F, Teitelbaum M, Orevi M, Horovitz A, Galun R. The saliva of the medicinal leech Hirudo medicinalis--II. Inhibition of platelet aggregation and of leukocyte activity and examination of reputed anaesthetic effects. Comp Biochem Physiol C Comp Pharmacol Toxicol. 1987;88(1):95-8. doi: 10.1016/0742-8413(87)90052-1. PMID 2890494
- [Background] Scott K. Is hirudin a potential therapeutic agent for arthritis? Ann Rheum Dis. 2002 Jun;61(6):561-2. doi: 10.1136/ard.61.6.561. No abstract available. PMID 12006337
- [Background] Bush D, Fritz H, Knight C, Mount J, Scott K. A hirudin-sensitive, growth-related proteinase from human fibroblasts. Biol Chem. 1998 Feb;379(2):225-9. doi: 10.1515/bchm.1998.379.2.225. PMID 9524076
- [Background] de Chalain TM. Exploring the use of the medicinal leech: a clinical risk-benefit analysis. J Reconstr Microsurg. 1996 Apr;12(3):165-72. doi: 10.1055/s-2007-1006471. PMID 8726336
- [Background] Lineaweaver WC, Hill MK, Buncke GM, Follansbee S, Buncke HJ, Wong RK, Manders EK, Grotting JC, Anthony J, Mathes SJ. Aeromonas hydrophila infections following use of medicinal leeches in replantation and flap surgery. Ann Plast Surg. 1992 Sep;29(3):238-44. doi: 10.1097/00000637-199209000-00008. PMID 1524373
- [Background] Fenollar F, Fournier PE, Legre R. Unusual case of Aeromonas sobria cellulitis associated with the use of leeches. Eur J Clin Microbiol Infect Dis. 1999 Jan;18(1):72-3. doi: 10.1007/s100960050232. No abstract available. PMID 10192721
- [Background] Ikizceli I, Avsarogullari L, Sozuer E, Yurumez Y, Akdur O. Bleeding due to a medicinal leech bite. Emerg Med J. 2005 Jun;22(6):458-60. doi: 10.1136/emj.2003.013847. PMID 15911965